CLINICAL TRIAL: NCT06383624
Title: Impact Of Maternal Spinal Anesthesia-Induced Hypotension At Scheduled Cesarean Delivery On Risk Development Of Transient Tachypnea Of Newborn And Fetal Acidosis: A Prospective Study
Brief Title: Impact Of Maternal Spinal Anesthesia-Induced Hypotension At Scheduled Cesarean Delivery On Risk Development Of Transient Tachypnea Of Newborn And Fetal Acidosis
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amany Mohammed El-Rebigi, MD, Lecturer of Pediatric and Neonatology, Benha University
Other Study IDs: RC18-4-2023
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Transient Tachypnea of Newborn and Fetal Acidosis
Keywords: Transient tachypnea of newborn, Fetal acidosis, Spinal anesthesia, Scheduled cesarean section
MeSH Terms: conditions — Transient Tachypnea of the Newborn

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We will evaluate the association between transient tachypnea of newborns and fetal acidosis development to the degree and duration of maternal hypotension and anesthesia to delivery time during spinal anesthesia at scheduled cesarean delivery.

DETAILED DESCRIPTION:
Transient tachypnea of the newborn (TTN) is characterized by mild to moderate respiratory distress that is a common self-limited disease of term newborns which gradually improves during the first 48 to 72 hours of life. TTN results from failure of the newborn to effectively clear the fetal lung fluid soon after birth.

It requires admission to the neonatal intensive care unit which leads to maternal-infant separation, the need for respiratory support, extended unnecessary exposure to antibiotics, prolonged hospital stays and increased health care costs.

Furthermore, these term neonates are at higher risk for inpatient admission for respiratory syncytial virus bronchiolitis in infancy and reactive airway disease later in life.

Transient tachypnea of newborns is 2- to 6-fold more common during elective cesarean delivery compared to vaginal birth.

Although the maternal-fetal risk factors for transient tachypnea of newborns are well understood, preoperative factors, especially in the setting of elective cesarean delivery, remain poorly investigated.

Significant maternal hypotension is a frequent complication of spinal anesthesia during caesarean delivery. However, spinal anesthesia is still the preferred anesthetic technique for cesarean delivery due to multiple factors such as avoiding risk of aspiration associated with general anesthetic, maternal ability to witness the birth of the baby and higher neonatal APGAR scores.

To our knowledge, no study has explored the potential role of maternal hemodynamic parameters during neuraxial anesthesia and effect of anesthesia to delivery time at scheduled cesarean delivery in the development of transient tachypnea of newborns and fetal acidosis in Egypt. Therefore, we hypothesized that pre-delivery maternal spinal anesthesia induced hypotension and anesthesia to delivery time would be associated with transient tachypnea of newborns and fetal acidosis in fullterm neonates delivered by elective cesarean section.

To test this hypothesis, we performed a prospective observational cohort study to evaluate the association of degree and duration of maternal hypotension and anesthesia to delivery time with development of transient tachypnea of newbon and fetal acidosis.

ELIGIBILITY:
Inclusion Criteria:

* Apparently normal singleton pregnancies with gestational age ≥37 weeks who will be underwent a scheduled elective cesarean section under spinal anesthesia.

Exclusion Criteria:

1. - Multiple pregnancies.
2. - Gestational age < 37 weeks.
3. - Neonates with congenital anomalies.
4. - Maternal exposure to antenatal steroids
5. - Mothers with medical problems as gestational or chronic diabetes mellitus and pregnancy induced hypertension or chronic hypertension.
6. - Induced or spontaneous onset of labor.
7. - Combined spinal-epidural anesthetic during which epidural activation is necessary before delivery .

Ages: 1 Minute to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All fullterm neonates born via scheduled cesarean delivery between April 2023 and March 2023 will be included in our study. All methods will be carried out in accordance with relevant guidelines and regulations.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Association between transient tachypnea of newborns development to the degree and duration of maternal hypotension during spinal anesthesia at scheduled cesarean delivery | 6 hours after delivery
  We will evaluate the association between transient tachypnea of newborns development to the degree and duration of maternal hypotension and anesthesia to delivery time during spinal anesthesia at scheduled cesarean delivery
Association between fetal acidosis development to the degree and duration of maternal hypotension and anesthesia to delivery time during spinal anesthesia at scheduled cesarean delivery | 1 hour after delivery
  we will evaluate the association between fetal acidosis development to the degree and duration of maternal hypotension and anesthesia to delivery time during spinal anesthesia at scheduled cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Amany M. El-Rebigi, MD, Principal Investigator — lecturer of pediatric and neonatology, Faculty of medicine, Benha University, Egypt
Locations (1):
- Benha University Hospital, Cairo, Egypt